CLINICAL TRIAL: NCT03678753
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Cenobamate Adjunctive Therapy in Subjects With PGTC Seizures
Brief Title: Randomized, Double-Blind Study to Evaluate Efficacy and Safety of Cenobamate Adjunctive Therapy in PGTC Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP3089C025
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Primary Generalized Epilepsy
Keywords: Primary Generalized Tonic-Clonic Seizures; PGTC; Idiopathic Generalized Epilepsy; Generalized Tonic-Clonic Seizures
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized; Seizures | interventions — Cenobamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenobamate (Experimental): Cenobamate 12.5 mg tablet once a day for two weeks, 25 mg tablet once a day for two weeks, 50 mg tablet once a day for two weeks, 100 mg tablets once a day for two weeks, 150 mg tablets once a day for two weeks and 200 mg tablets once a day for twelve weeks. Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight.
  Interventions: Drug: Cenobamate
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenobamate — 12.5 mg tablet, 25 mg tablet, 50 mg tablet, 100 mg tablets, 150 mg tablets, 200 mg tablets. Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight.
  Other Names: YKP3089
  Arms: Cenobamate
Drug: Placebo — Matching Placebo
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This trial is intended to study the safety and effectiveness of an new anti-epileptic drug (AED) on Primary Generalized Tonic-Clonic (PGTC) Seizures. Eligible Subjects, adults and adolescents, will continue to take their usual AEDs and receive either cenobamate or placebo. Subjects will have a 50% chance or receiving cenobamate or placebo (sugar pill). Subjects will initially receive 12.5 mg of cenobamate or placebo (study drug) and increase the dose every two weeks until they reach a target dose of 200 mg. Subjects will take study drug at approximately the same time in the morning (once a day) with or without food. If tolerability issues arise, dosing can be changed to evening. Also, once a subject reaches 200 mg, the dose can be decreased one time to 150 mg, if necessary. The treatment period is 22 weeks and there is a 3 week follow up period, which includes a one week decrease in study drug to 100 mg prior to stopping. Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight. Subjects who complete may be eligible for an extension study and will not have to complete the follow up period. Subjects will track their seizure types and frequency in a diary throughout the study.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo controlled trial is designed to evaluate safety, efficacy, and pharmacokinetics of cenobamate adjunctive therapy as compared to placebo on PGTC seizures in subject with idiopathic generalized epilepsy. Subjects will be randomized to receive either cenobamate or placebo on a 1:1 basis. The study will have three periods, pre-randomization period where a baseline seizure frequency is established, treatment period and follow up period. The treatment period consists of a 10 week titration phase where subjects are titrated slowly until they reach the target dose and a maintenance phase. During the titration phase, subjects will receive 12.5 mg study drug, followed by 25 mg, 50 mg, 100 mg, and 150 mg study drug every two weeks. During the maintenance phase, subjects will receive the target dose of 200 mg study drug or adolescent equivalent. Subjects will take their once daily dose of study drug at approximately the same in the morning with or without food. If tolerability issues arise, subjects can switch to evening dosing. There is also an option to down-titrate to 150 mg study drug, one time only. If tolerability issues continue, subjects may be discontinued. Upon completion of the maintenance phase, eligible subjects will have an opportunity to enroll in an open-label safety study. Subjects who discontinue early or do not wish to participate in this additional study will complete the three week follow up period. Subjects may receive a one week down titration to 100 mg and return for a follow up visit 2 weeks later. Adolescents will follow the same every two week regimen and receive cenobamate as an oral suspension based on weight Throughout the study, subjects will keep a diary containing the type and frequency of seizures. This will be the primary efficacy measure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female and aged ≥12 years.
2. Written informed consent signed by the subject or legal guardian, or legally authorized representative (LAR), prior to entering the study, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines. Age- appropriate assent will be obtained for adolescents. If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained. As required by country-specific regulations, only the subject may sign the Informed Consent Form (ICF) in accordance with ICH guidelines.
3. Female subjects of childbearing potential are willing to use an acceptable form of birth control
4. Subject has a clinical diagnosis of PGTC seizures (with or without other subtypes of generalized seizures) in the setting of idiopathic generalized epilepsy.
5. Subject experiences at least 5 PGTC seizures in 12 weeks during the Pre-Randomization Period.
6. Subject has had a routine electroencephalogram (EEG) within 5 years prior to Visit1 (Screening/Baseline) or during the Pre-Randomization Period with electroencephalographic features consistent with idiopathic generalized epilepsy; other concomitant anomalies must be explained by adequate past medical history.
7. Subject has undergone computed tomography (CT) or magnetic resonance imaging (MRI) within 10 years prior to Visit 1 (Screening/Baseline) or during the Pre-Randomization Period that ruled out a progressive cause of epilepsy.
8. Subject is currently receiving 1 to a maximum of 3 concomitant AEDs with fixed dosing regimens for a minimum of 30 days prior to Visit 1 (Screening/Baseline).

   1. Benzodiazepines (except diazepam, see Exclusion Criterion No.7) taken at least once per week during the 30 days prior to Visit 1 (Screening/Baseline) for epilepsy, anxiety, or sleep disorder will be counted as 1 AED and the dosage must be continued unchanged throughout the study. Therefore, only a maximum of 2 additional approved AEDs will be allowed. (See Exclusion Criterion No. 10 for intermittent benzodiazepine rescue parameters.)
   2. Subjects receiving felbamate as a concomitant AED must meet the following criteria: i. Have a 2-year history of felbamate use and a history of a fixed dosing regimen for a minimum of 60 days prior to Visit 1 (Screening/Baseline). ii. No prior or known history of hepatotoxicity or hematologic disorder due to felbamate.
9. Subject with an implanted vagal nerve or deep brain stimulator will be allowed if the stimulator was implanted at least 5 months prior to Visit 1 (Screening/Baseline) and the stimulator parameters are not changed for 30 days prior to Visit 1 and for the duration of the study.
10. Subject taking a ketogenic diet will be allowed as long as the diet has been stable for at least 3 months prior to Visit 1 (Screening/Baseline) and will remain stable for the duration of the study.

Exclusion Criteria:

1. Female subjects who are pregnant (or planning to become pregnant during the study), lactating, or breast-feeding.
2. Subject has a history o f status epilepticus that required hospitalization within 12 months prior to Visit 1 (Screening/Baseline).
3. Subject has PGTC seizure clusters where individual seizures cannot be counted or classified.
4. Subject has a history of non-epileptic psychogenic seizures.
5. Subject has a concomitant diagnosis of Partial Onset Seizures (POS).
6. Subject has a clinical diagnosis of Lennox-Gastaut syndrome.
7. Subject is currently taking (within the 30 days prior to Visit 1 [Screening/Baseline]) any of the following medications: diazepam (for any reason other than as intermittent benzodiazepine rescue medication), phenytoin, mephenytoin, fosphenytoin, phenobarbital, primidone, ethotoin, clopidogrel, fluvoxamine, amitriptyline, clomipramine, bupropion, methadone, ifosfamide, cyclophosphamide, or efavirenz.
8. Subject has participated in previous cenobamate clinical studies.
9. Subject has a history of vigabatrin use within 5months prior to Visit 1 (Screening/Baseline), or the subject plans to begin treatment with vigabatrin during the study.

   a) A subject with a history of vigabatrin use that ended more than 5 months prior to Visit1 may be enrolled after documented evidence of no vigabatrin-associated clinically significant abnormality in an automated visual perimetry test.
10. Subject has a history of intermittent use of rescue benzodiazepines (i.e., 1 to 2 doses over a 24-hour period is considered a 1-time rescue) 4 or more times within the 30 days prior to Visit 1 (Screening/Baseline).
11. Subject has received an investigational drug or device within 30 days prior to Visit 1 (Screening/Baseline).
12. Subject has a history of drug or alcohol dependency or abuse within 2 years prior to Visit 1 (Screening/Baseline).
13. Subject tests positive, via urine drug screen at Visit 1 (Screening/Baseline), for illicit drugs not legalized in your region/state, or for a drug that has not been prescribed (e.g., certain opiates).
14. Subject has a history of any serious drug-induced hypersensitivity reaction (including, but not limited to, Stevens Johnson syndrome, toxic epidermal necrolysis, or DRESS) or any drug-related rash requiring hospitalization.
15. History of AED-associated rash that involved conjunctiva or mucosae.
16. History of more than one non-serious drug-related hypersensitivity reaction that required discontinuation of the medication.
17. Subject has evidence of clinically significant abnormalities or disease (e.g., psychiatric, cardiac, respiratory, gastrointestinal, hepatic [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 2 times the upper limit of normal (ULN), or total or direct bilirubin not more than ULN], or renal disease) that, in the opinion of the Principal Investigator, could affect the subject's safety or conduct of the study.
18. Presence of congenital short QT syndrome or relevant replicated change in QT/QTc interval less than 340 msec on ECG.
19. Subject has any significant active Central Nervous System (CNS) infection, demyelinating disease, degenerative neurologic disease or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results.
20. Subject has a creatinine clearance less than 50 mL/min, as calculated by Cockcroft-Gault equation.
21. Subject has an absolute neutrophil count less than 1500/µL.
22. Subject has platelet count lower than 80,000/µL in subjects treated with valproate.
23. Subject has a history of positive antibody/antigen test for hepatitis A, hepatitis B, hepatitis C, or HIV.
24. Subject has any suicidal ideation (with intent with or without a plan) at Visit 1 (Screening/Baseline) or Visit 4 (Randomization) (i.e., answering YES to Question 4 and/or Question 5 on the Suicidal Ideation section of the C-SSRS).
25. Subject has more than 1 lifetime suicide attempt.
26. Subject is a staff member or immediate family member of study staff.
27. Previous exposure to cenobamate or sensitivity/allergy to components of the oral suspension.

Any potential exception to the inclusion as well as exclusion criteria allowing de minimis (clinically trivial and meaningless) variations must be approved by the Medical Monitor.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Seizure Diary | 28 Days
  Daily seizure diary that contains type and frequency of seizures

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Misra, MD, Study Director — SK Life Science, Inc.
Locations (116):
- United States (43):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Neuro Pain Medical Center, Fresno, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Children's Hospital of Colorado, Grand Junction, Colorado
  - Brainstorm Research, Miami, Florida
  - Florida Hospital Medical Group, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Clinical Integrative Research Center of Atlanta, CIRCA, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, Boise, Idaho
  - Rush University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - PMG Research of McFarland Clinic, Ames, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic of Neurology Golden Valley, Golden Valley, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - JFK Medical Center- The Neuroscience Institute, Edison, New Jersey
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - New York Presbyterian Hospital, Brooklyn, New York
  - UBMD Neurology, Buffalo, New York
  - Five Towns Neuroscience Research, Woodmere, New York
  - Duke University Children's Health Center, Durham, North Carolina
  - Ohio Health Research and Innovation Institute, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Child Neurology Consultants of Austin, Austin, Texas
  - ANRC Research, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah / Primary Children's Hospital, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
  - Valley Medical Center, Renton, Washington
  - MultiCare Institute for Research and Innovation, Spokane, Washington
- Australia (2):
  - Austin Health, Heidelberg
  - Children's Health Queensland Hospital, South Brisbane
- Bulgaria (8):
  - MHAT Sv. Ivan Rilski Gorna Oryahovitsa EOOD, Gorna Oryahovitsa, Veliko Tarnovo
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - UMHAT Kanev AD, Rousse
  - MHAT Lyulin EAD, Sofia
  - Acibadem City Clinic MHAT Tokuda EAD, Sofia
  - Diagnostic Consultative Center Neoclinic EAD, Sofia
  - Diagnostic Consultative Center Equita EOOD, Varna
  - Medical Center Medica Plus OOD, Veliko Tarnovo
- Czechia (8):
  - Fakultní nemocnice v Motole, Prague, Prague
  - Fakultni nemocnice u sv. Anny v Brne, 1. Neurologicka klinika, Brno
  - Nestatni zdravotnicke zarizeni, privatni ordinance neurologie, Hradec Králové
  - Cerebrovaskularni poradna, s.r.o., Ostrava-Poruba
  - Cerebovaskularni poradna s.r.o., Ostrava-Vitkovice
  - Forbeli s.r.o., Neurologicka ordinace, Prague
  - Vestra Clinics, s.r.o., Rychnov nad Kněžnou
  - Neurologicka ambulance MUDr.Monika Zahumenska, Zlín
- Georgia (2):
  - LEPL Tbilisi State Medical University Givi Zhvania Academic Clinic of Pediatry, Tbilisi
  - Institute of Neurology and Neuropsychology LTD, Tbilisi
- Germany (4):
  - Charite - Universitätsmedizin Berlin - Sozialpädiatrisches Zentrum, Berlin
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Sächsisches Epilepsiezentrum Kleinwachau gGmbH, Radeberg
- Hungary (3):
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Központ, Gyermekgyógyászati Intézet Nagyerdei krt. 98, Debrecen
  - Csongrád Megyei Egészségügyi Elláto Központ Ideggyógyászati Osztály, Hódmezővásárhely
- Poland (16):
  - Clinical Research Center Spolka z Ograniczona Odpowiedzialnoscia Medic-R sp. k, Poznan, Greater Poland Voivodeship
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska S.J., Ksawerów, Iodzkie
  - Centrum Leczenia Padaczki i Migreny, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Plejady, Krakow, Lesser Poland Voivodeship
  - Wojewódzki Specjalistyczny Szpital Dziecięcy im. sw. Ludwika sw Krakowie, Krakow, Lesser Poland Voivodeship
  - NZOZ Poradnia Zdrowia Psychicznego Antonijczuk Boleslaw, Tyniec Mały, Lower Silesian Voivodeship
  - Centrum Medyczne Oporów, Wroclaw, Lower Silesian Voivodeship
  - Instytut Medycyny Wsi im. Witolda Chodzki w Lublinie, Lublin, Lublin Voivodeship
  - Centrum Medyczne Warszawa Pratia s.a, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Pratia Katowice, Katowice, Silesian Voivodeship
  - M.A. LEK A.M. Maciejowscy S.C Centrum Terapii SM, Katowice, Silesian Voivodeship
  - Gornoslaskie Centrum Medyczne - Samodzielny Publiczny Szpital Kliniczny Number 7, Katowice, Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Novo-Med, Katowice, Silesian Voivodeship
  - Gyncentrum Clinic Sp. z.o.o, Katowice, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej - Centrum Neurologii Dziecięcej i Leczenia Padaczki, Kielce, Świętokrzyskie Voivodeship
- Slovakia (6):
  - Konzílium, s.r.o, Dubnica nad Váhom, Trenčín Region
  - MUDr. Beata Dupejova, neurologická ambulncia, s.r.o, Banská Bystrica
  - IN MEDIC s.r.o, Bardejov
  - Narodny Ustav Detskych Chorob, Bratislava
  - MEDBAJ, s.r.o., Neurologicka ambulancia, Nemocnicna 1944/10, Dolný Kubín
  - NEURES, s.r.o.-Neurologická Ambulancia, Krompachy
- South Korea (4):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - SMG-SNU Boramae Medical Center, Seoul, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Ajou University Hospital, Suwon
- Spain (3):
  - Hospital Clínico San Carlos, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario La Fe, Valencia
- Ukraine (17):
  - Municipal Non-profit Enterprise City Clinical Hospital No.16 of Dnipro City Council, Department of Neurology, Dnipro, Dnipropetrovsk Oblast
  - Communal Enterprise Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnykov of Dnipropetrovsk Regional Council, Regional Center of Psychosomatic Disorders based on Psychoneurology Department, Dnipro, Dnipro
  - Kyiv City Psychoneurological Hospital №2, Kiev, Kyiv Oblast
  - Municipal Non-Profit Enterprise Odesa Regional Clinical Hospital of Odesa Regional Council, Department of Cerebro-Vascular Diseases with Neurosurgery, Odesa, Odesa Oblast
  - Municipal Non-profit Enterprise Regional Clinical Center of Neurosurgery and Neurology of Zakarpattia Regional Council, Department of Neurosurgery #2, Uzhhorod, Zakarpattia Oblast
  - Municipal Non-Profit Enterprise Zaporizhzhia Regional Clinical Hospital Of Zaporizhzhia Regional Council, Zaporizhzhya, Zaporizhzhya
  - Communal Enterprise Regional Medical Center of Family Health of the Dnipropetrovsk Regional Council, Dnipro
  - Communal Non-commercial Enterprise City Children's Clinical Hospital 6 of Dnipro City Council, Dnipro
  - Communal Enterprise Dnipropetrovsk Regional Clinical Hospital n.a. I.I. Mechnykov of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - Municipal Non-profit Enterprise Prykarpattia Regional Clinical Center for Mental Health of Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Communal Non-Commercial Enterprise of Kharkiv Regional Council Regional Clinical Psychiatric Hospital #3, Kharkiv
  - Communal Non-Profit Enterprise of Lviv Regional Council Lviv Regional Clinical Hospital, Neurological Department, Antiepileptic Center, Lviv
  - Communal Non-Profit Enterprise Odesa Regional Medical Centre of Mental Health Odesa Regional Council, Department #2, Odesa
  - Odessa Regional Psychiatric Hospital No. 2,, Odesa
  - Communal Enterprise Poltava Regional Clinical Psychiatric Hospital named after O.F. Maltsev of Poltava Regional Council, Poltava
  - Municipal Non-Profit Enterprise Ternopil Regional Clinical Psychoneurological Hospital of Ternopil Regional Council, Department of Neurology #2, Ternopil
  - Municipal Non-profit Enterprise Vinnytsia Regional Clinical Psychoneurological Hospital named after Acad. O.I. Yushchenko of Vinnytsia Regional Council, Department of Neurology #3, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brigo F, Lattanzi S. Cenobamate add-on therapy for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2024 Aug 1;8(8):CD014941. doi: 10.1002/14651858.CD014941.pub2. PMID 39087564
- [Derived] Rosenfeld WE, Ferrari L, Kamin M. Efficacy of cenobamate by focal seizure subtypes: Post-hoc analysis of a phase 3, multicenter, open-label study. Epilepsy Res. 2022 Jul;183:106940. doi: 10.1016/j.eplepsyres.2022.106940. Epub 2022 May 5. PMID 35605481